CLINICAL TRIAL: NCT03501082
Title: Rewilding the Human Gut: Reintroduction of the Species Limosilactobacillus Reuteri
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: Pro00077565
Record Dates: First submitted 2017-11-21; First posted 2018-04-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-05

CONDITIONS: Microbial Colonization
Keywords: Gut microbiome
MeSH Terms: conditions — Communicable Diseases | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Crossover design for dietary intervention (non-industrialized-type diet compared to participants' usual diet); parallel design for L. reuteri probiotic (L. reuteri PB-W1, L. reuteri DSM-20016T, and placebo).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- L. reuteri PB-W1, Non-Industrialized-Type Diet Start (Experimental): Participants will receive the non-industrialized-type diet for 3 weeks, followed by a crossover to 3 weeks of consuming their usual diet after a 3-week washout period. Participants will be provided with a one-time dose of L. reuteri PB-W1 strain on day 4 of each diet period. The L. reuteri PB-W1 strain will be provided as a drinkable solution (approximately 2.25x10^10 viable cells will be provided in 50 ml of water).
  Interventions: Other: L Reuteri PB-W1 Strain; Other: Non-Industrialized-Type Diet
- L. reuteri DSM20016T, Non-Industrialized-Type Diet Start (Experimental): Participants will receive the non-industrialized-type diet for 3 weeks, followed by a crossover to 3 weeks of consuming their usual diet after a 3-week washout period. Participants will be provided with a one-time dose of L. reuteri DSM20016T strain on day 4 of each diet period. The L. reuteri DSM20016T strain will be provided as a drinkable solution (approximately 2.25x10^10 viable cells will be provided in 50 ml of water).
  Interventions: Other: L. Reuteri DSM20016T Strain; Other: Non-Industrialized-Type Diet
- Placebo, Non-Industrialized-Type Diet Start (Placebo Comparator): Participants will receive the non-industrialized-type diet for 3 weeks, followed by a crossover to 3 weeks of consuming their usual diet after a 3-week washout period. Participants will be provided with a one-time dose of a placebo solution on day 4 of each diet period. The placebo solution will be provided as a drinkable solution (2 g maltodextrin dissolved in 50 ml water in food grade conditions).
  Interventions: Other: Placebo; Other: Non-Industrialized-Type Diet
- L. reuteri PB-W1, Usual Diet Start (Experimental): Participants will consume their usual diet for 3 weeks, followed by a crossover to 3 weeks of consuming the provided non-industrialized-type diet after a 3-week washout period. Participants will be provided with a one-time dose of L. reuteri PB-W1 strain on day 4 of each diet period. The L. reuteri PB-W1 strain will be provided as a drinkable solution (approximately 2.25x10^10 viable cells will be provided in 50 ml of water).
  Interventions: Other: L Reuteri PB-W1 Strain; Other: Non-Industrialized-Type Diet
- L. reuteri DSM20016T, Usual Diet Start (Experimental): Participants will consume their usual diet for 3 weeks, followed by a crossover to 3 weeks of consuming the provided non-industrialized-type diet after a 3-week washout period. Participants will be provided with a one-time dose of L. reuteri DSM20016T strain on day 4 of each diet period. The L. reuteri DSM20016T strain will be provided as a drinkable solution (approximately 2.25x10^10 viable cells will be provided in 50 ml of water).
  Interventions: Other: L. Reuteri DSM20016T Strain; Other: Non-Industrialized-Type Diet
- Placebo, Usual Diet Start (Placebo Comparator): Participants will consume their usual diet for 3 weeks, followed by a crossover to 3 weeks of consuming the provided non-industrialized-type diet after a 3-week washout period. Participants will be provided with a one-time dose of a placebo solution on day 4 of each diet period. The placebo solution will be provided as a drinkable solution (2 g maltodextrin dissolved in 50 ml water in food grade conditions).
  Interventions: Other: Placebo; Other: Non-Industrialized-Type Diet

INTERVENTIONS:
Other: L Reuteri PB-W1 Strain — L. Reuteri PB-W1 strain will be prepared in accordance to the standardized operating procedures to prepare Limosilactobacillus reuteri in food grade conditions
  Other Names: Probiotic
  Arms: L. reuteri PB-W1, Non-Industrialized-Type Diet Start; L. reuteri PB-W1, Usual Diet Start
Other: L. Reuteri DSM20016T Strain — L. Reuteri DSM20016T strain will be prepared in accordance to the standardized operating procedures to prepare Limosilactobacillus reuteri in food grade conditions
  Other Names: Probiotic
  Arms: L. reuteri DSM20016T, Non-Industrialized-Type Diet Start; L. reuteri DSM20016T, Usual Diet Start
Other: Placebo — 2 g of maltodextrin will be dissolved in 50 ml water in food grade conditions
  Arms: Placebo, Non-Industrialized-Type Diet Start; Placebo, Usual Diet Start
Other: Non-Industrialized-Type Diet — Non-industrialized-type diet will be prepared in a metabolic kitchen, with all meals and snacks provided to participants for three weeks.
  Other Names: Controlled Diet

SUMMARY:
The large intestine is home to trillions of microbes, known as the gut microbiome, which perform essential functions, such as digesting food and fighting disease. The diversity of microbes present in our gut microbiome is influenced by lifestyle factors, such as dietary patterns, medication usage, and sanitation practices. Research shows that the diversity of the human gut microbiome decreases as societies undergo industrialization. For example, fecal samples from rural Papua New Guineans contain an additional 50 microbial species, such as Limosilactobacillus reuteri, not found in people living in the United States.

What has caused the disappearance of L. reuteri in industrialized countries is currently unknown. However, diet is a major factor influencing the composition of the gut microbiome. Microbiota-accessible carbohydrates (MACs) are indigestible carbohydrates that are a primary source of energy for gut microbes. North Americans consume far less of these carbohydrates (which are contained in foods such as beans, yams, and artichokes) than rural Papua New Guineans.

The overall aim of this controlled feeding study is to determine if a strain of L. reuteri isolated from rural Papua New Guinea can be established in the gut of Canadians when taken as a probiotic alongside a non-industrialized-type diet designed to promote its growth. Furthermore, the study will determine:

(i) the physiological and immunological effects of both L. reuteri and the non-industrialized-type diet, and (ii) the effects of both L. reuteri and the non-industrialized-type diet on gut microbiome ecology.

DETAILED DESCRIPTION:
There is now consistent evidence that industrialization has substantially decreased the bacterial diversity of the gut microbiota (Segata, 2015), likely due to a combination of factors such as use of antibiotics, modern clinical practices, sanitation, and changes in dietary habits. However, the only factor for which empirical evidence exists is the low content of Microbiota-Accessible Carbohydrates (MACs) in Western diets, which are indigestible dietary carbohydrates that become available to the microbes colonizing the intestine (Sonnerburg et al., 2015).

Previous work has confirmed the overall premise of 'microbiome depletion' by demonstrating higher diversity in the fecal microbiota of individuals from rural tribes in Papua New Guinea, which contain an additional of 50 species completely undetectable in North Americans (Martínez et al., 2015). One species detectable in every Papua New Guinean individual by 16S rRNA sequencing but not in a single US control was Limosilactobacillus reuteri (L. reuteri). Interestingly, this species, which is also used as a probiotic, was regularly detected in humans in studies conducted around 1960, but is very rarely found in contemporary humans, suggesting a recent decline of the L. reuteri population in Westerners (Walter et al., 2011). Most importantly, L. reuteri is a member of the gut microbiota in many vertebrate species and exerts benefits towards host immune functions and development, as demonstrated in a number of highly cited publications (Zelante et al. 2013; Buffington et al. 2016; Lamas et al. 2016; He et al. 2017).

It is currently unclear what caused the drop in the L. reuteri population. However, it is likely due to the importance of non-digestible carbohydrates that are present at very low amounts in Western diets, while being abundant in the diet of rural Papua New Guineans, a population that consumes a predominantly plant-based diet.

The goal of this study is to demonstrate that a bacterial species dominant in the non-westernized microbiome can be 'reintroduced' in the gut of Canadians fed a non-industrialized type diet designed to promote the growth of gut bacteria. This study will also determine how this 'reintroduction' and the non-industrialized-type diet influences immune function of the host and host-diet-microbiome metabolic interactions, and explore associations between them. It will further explore the effects of the microbial treatment and the diet on gut microbiome ecology. The central hypothesis is that an isolate of L. reuteri, originating from rural Papua New Guinea, can be established in the gut of Canadians fed a diet containing the carbohydrates known to facilitate the growth of this microbe. It is also hypothesized that this 'reintroduction' and consuming the non-industrialized type diet will be associated with immunological and metabolic benefits to the host. To achieve these goals, the following aims are proposed:

1. To conduct a human trial to determine if a Limosilactobacillus reuteri strain isolated from rural Papua New Guinea (PNG) can be established in the gut of healthy Canadians.
2. To determine if colonization can be improved by feeding a diet specifically designed to provide growth substrates for L. reuteri.
3. To determine how both L. reuteri and the non-industrialized-type diet change the human microbiome, metabolome, cardiometabolic surrogate endpoints, and immune biomarkers of inflammation.

This study will establish if a 'lost species' of bacteria can be reintroduced into the human gut and may provide mechanistic insight to inform how such dietary modulation may be applied to reduce the risk of chronic diseases. Since the L. reuteri strain isolated from rural Papua New Guineans is functionally different from western strains, evidenced by different growth rates on substrates of MACs, this study will further identify potential probiotic strains that were previously uncharacterized due to their overall absence from the industrialized gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals with a body mass index between 20-29.9 kg/m²
* Have at least one bowel movement per day
* Willing to consume prepared study foods (breakfast, lunch dinner, snacks) for a period of 3 weeks
* Men and pre-menopausal, non-pregnant or non-lactating women
* Non-vegetarian, non-smoking, and alcohol intake ≤8 drinks/week, and willing to consume 8 drinks per week or less during the course of the study.
* If consuming probiotic containing foods, willing to discontinue eating same, and substitute with non-probiotic containing foods

  -≤5 h/week of moderate-vigorous exercise.
* Quantity of L. reuteri in screening fecal sample below 10^4 CFU/g

Exclusion Criteria:

* History of diabetes, acute or chronic GI illnesses, conditions, or history of GI surgical intervention
* antibiotic treatment in the last 3 months
* use of dietary supplements (including prebiotics and probiotics, fiber supplements/bars, digestive enzymes/beano)- if consumed, willing to undergo 4 week pre-intervention washout period, and remain free of supplements for duration of study. Exception: multivitamin or vitamin d supplement (1 week washout period)
* use of antihypertensive, lipid-lowering, anti-diabetic, anti-inflammatory (i.e corticosteroids or chronic NSAID use), or laxative medications
* known food allergies or intolerances (including dairy allergic or lactose intolerant)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Establishment of L. reuteri (PB-W1 & DSM20016T strains) in the gut of Canadian individuals | 21 days
  The primary outcome of this study is to measure L. reuteri (PB-W1 and DSM20016T strains) establishment in the gut of Canadian individuals. This will be measured by selective bacterial culture from fecal samples and quantified through quantitative PCR using species specific primers.
Enhanced persistence of colonization of L. reuteri (PB-W1 & DSM20016T strains) following consumption of non-industrialized-type diet designed to provide growth substrates for L. reuteri | 21 days
  We will measure if the persistence of L. reuteri in the gut of Canadian individuals is enhanced by the consumption of a non-industrialized-type diet specifically designed to provide growth substrates (MACs) for L. reuteri. This will be measured by selective bacterial culture from fecal samples and quantified through quantitative PCR using species specific primers.

SECONDARY OUTCOMES:
Effect of L. reuteri strains and the non-industrialized-type diet on cardiometabolic surrogate endpoints: fasting glucose and lipid panel. | 21 days
  Plasma from blood samples will be analyzed for changes in glucose, triglycerides, low density lipoprotein (LDL) cholesterol, high density lipoprotein (HDL) cholesterol, non-HDL cholesterol, and total cholesterol (mmol/L).
Effect of L. reuteri strains and the non-industrialized-type diet on cardiometabolic surrogate endpoints: fasting insulin levels. | 21 Days
  Plasma from blood samples will be analyzed for changes in insulin (µIU/L).
Effect of L. reuteri strains and the non-industrialized-type diet on cardiometabolic surrogate endpoints: homeostatic model assessment of insulin resistance and quantitative insulin sensitivity check index. | 21 Days
  Homeostatic model assessment of insulin resistance and quantitative insulin sensitivity check index will be calculated based on fasting glucose and insulin levels.
Effect of L. reuteri strains and the non-industrialized-type diet on cardiometabolic surrogate endpoints: fasting C-reactive protein levels. | 21 Days
  Plasma from blood samples will be analyzed for changes in C-reactive protein (mg/L).
Effect of L. reuteri strains and the non-industrialized-type diet on cardiometabolic surrogate endpoints: body weight. | 21 Days
  Body weight will be measured in kilograms.
Effect of L. reuteri strains and the non-industrialized-type diet on inflammatory bowel disease surrogate endpoint: fecal calprotectin levels. | 21 Days
  Fecal samples will be analyzed for changes in calprotectin (ng/mg).
Effect of L. reuteri strains and the non-industrialized-type diet on biomarkers of gut barrier function: lipopolysaccharide binding protein. | 21 Days
  Plasma from blood samples will be analyzed for changes in lipopolysaccharide binding protein (µg/mL).
Effect of L. reuteri strains and the non-industrialized-type diet on biomarkers of gut barrier function: fecal zonulin levels. | 21 days
  Fecal samples will be analyzed for changes in zonulin (ng/mg).
Effect of L reuteri strains and the non-industrialized-type diet on the composition of the fecal microbiome. | 4-21 days
  o Fecal samples will be analyzed using 16S rRNA-sequencing to measure changes in the fecal microbiome at the phylum, class, order, family, genus, and amplicon sequencing variant levels. Fecal microbiome composition will also be analyzed using whole metagenome sequencing to measure changes at the phylum, class, order, family, genus, species, and species-level genome bin levels.
Effect of L reuteri strains and the non-industrialized-type diet on the function of the fecal microbiome: enzyme levels. | 8 days
  Fecal samples will be analyzed using whole metagenome sequencing to measure changes in enzymes encoded by gut microbiota.
Effect of L reuteri strains and the non-industrialized-type diet on the function of the fecal microbiome: short-chain fatty acid levels. | 8 & 21 days
  Short-chain fatty acids (acetate, propionate, butyrate, valerate) and branched-chain fatty acids (isovalerate, isobutyrate) will be measured in fecal samples using gas chromatography mass spectrometry (µmol/g).
Effect of L reuteri strains and the non-industrialized-type diet on the function of the fecal microbiome: pH. | 8 & 21 days
  Fecal pH will be measured using a pH meter.
Effect of L. reuteri strains and non-industrialized-type diet on the metabolome. | 8 & 21 days
  Plasma metabolome will be assessed to determine changes in molecules with known immunological functions such as indole derivatives of tryptophan and bile acids following the provision of the intervention. This will be measured via high performance chemical isotope labeling liquid chromatography mass spectrometry platform.
Effect of L. reuteri strains and the non-industrialized-type diet on host immune response. | 8 & 21 days
  Host immune responses will be measured in blood samples by quantifying IgA, selected cytokines, and white blood cell phenotyping using flow cytometry. Mononuclear cells will be isolated from whole blood on ficoll gradients and the ability of cells to respond to challenges (peptidoglycan, phytohemagglutinin, and lipopolysaccharide) will be determined ex vivo.
Effect of L. reuteri strains and the non-industrialized-type diet on changes in psychological mood state. | 21 days
  Changes in individual mood state will be measured by the profile of mood states questionnaire (scored between -32 and 200; lower scores indicate more stable mood profiles).
Effect of L. reuteri strains and the non-industrialized-type diet on changes in gastrointestinal symptoms. | 21 days
  Changes in individual gastrointestinal symptoms will be measured by a gastrointestinal symptom questionnaire (scored on a scale of 0-5; higher scores indicating more symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Jens Walter, PhD, Principal Investigator — University College Cork; Andrea Haqq, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared that underlies the results reported after deidentification (text, tables, figures, and appendices). Data will be made available through a safe and secure publicly available data sharing repository.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication, ending 5 years following publication.
Access Criteria: Anyone who wishes to access the data may do so to achieve aims in the approved proposal and for individual participant data meta-analysis.

REFERENCES:
- [Background] Segata N. Gut Microbiome: Westernization and the Disappearance of Intestinal Diversity. Curr Biol. 2015 Jul 20;25(14):R611-3. doi: 10.1016/j.cub.2015.05.040. PMID 26196489
- [Background] Sonnenburg ED, Sonnenburg JL. Starving our microbial self: the deleterious consequences of a diet deficient in microbiota-accessible carbohydrates. Cell Metab. 2014 Nov 4;20(5):779-786. doi: 10.1016/j.cmet.2014.07.003. Epub 2014 Aug 21. PMID 25156449
- [Background] Martinez I, Stegen JC, Maldonado-Gomez MX, Eren AM, Siba PM, Greenhill AR, Walter J. The gut microbiota of rural papua new guineans: composition, diversity patterns, and ecological processes. Cell Rep. 2015 Apr 28;11(4):527-38. doi: 10.1016/j.celrep.2015.03.049. Epub 2015 Apr 16. PMID 25892234
- [Background] Walter J, Britton RA, Roos S. Host-microbial symbiosis in the vertebrate gastrointestinal tract and the Lactobacillus reuteri paradigm. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4645-52. doi: 10.1073/pnas.1000099107. Epub 2010 Jun 25. PMID 20615995
- [Background] Zelante T, Iannitti RG, Cunha C, De Luca A, Giovannini G, Pieraccini G, Zecchi R, D'Angelo C, Massi-Benedetti C, Fallarino F, Carvalho A, Puccetti P, Romani L. Tryptophan catabolites from microbiota engage aryl hydrocarbon receptor and balance mucosal reactivity via interleukin-22. Immunity. 2013 Aug 22;39(2):372-85. doi: 10.1016/j.immuni.2013.08.003. PMID 23973224
- [Background] Buffington SA, Di Prisco GV, Auchtung TA, Ajami NJ, Petrosino JF, Costa-Mattioli M. Microbial Reconstitution Reverses Maternal Diet-Induced Social and Synaptic Deficits in Offspring. Cell. 2016 Jun 16;165(7):1762-1775. doi: 10.1016/j.cell.2016.06.001. PMID 27315483
- [Background] Lamas B, Richard ML, Leducq V, Pham HP, Michel ML, Da Costa G, Bridonneau C, Jegou S, Hoffmann TW, Natividad JM, Brot L, Taleb S, Couturier-Maillard A, Nion-Larmurier I, Merabtene F, Seksik P, Bourrier A, Cosnes J, Ryffel B, Beaugerie L, Launay JM, Langella P, Xavier RJ, Sokol H. CARD9 impacts colitis by altering gut microbiota metabolism of tryptophan into aryl hydrocarbon receptor ligands. Nat Med. 2016 Jun;22(6):598-605. doi: 10.1038/nm.4102. Epub 2016 May 9. PMID 27158904
- [Background] He B, Hoang TK, Wang T, Ferris M, Taylor CM, Tian X, Luo M, Tran DQ, Zhou J, Tatevian N, Luo F, Molina JG, Blackburn MR, Gomez TH, Roos S, Rhoads JM, Liu Y. Resetting microbiota by Lactobacillus reuteri inhibits T reg deficiency-induced autoimmunity via adenosine A2A receptors. J Exp Med. 2017 Jan;214(1):107-123. doi: 10.1084/jem.20160961. Epub 2016 Dec 19. PMID 27994068